CLINICAL TRIAL: NCT00923260
Title: Effect of Omentectomy on Metabolic Syndrome, Acute Phase Reactants & Inflammatory Mediators in Patients Undergoing LRYGBP: A Randomized Trial
Brief Title: Omentectomy and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Miguel Francisco Herrera, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCMNSZ-1486
Record Dates: First submitted 2009-01-28; First posted 2009-06-18 (Estimated); Results first posted 2009-06-18 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-11

CONDITIONS: Metabolic Syndrome; Morbid Obesity
Keywords: Omentectomy; metabolic syndrome; acute phase reactants
MeSH Terms: conditions — Metabolic Syndrome; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roux-en-Y Gastric Bypass/Omentectomy (Experimental): Laparoscopic Roux-en-Y Gastric Bypass with omentectomy
  Interventions: Procedure: Laparoscopic Roux-en-Y Gastric Bypass; Procedure: Omentectomy
- Roux-en-Y Gastric Bypass alone (Active Comparator)
  Interventions: Procedure: Laparoscopic Roux-en-Y Gastric Bypass

INTERVENTIONS:
Procedure: Laparoscopic Roux-en-Y Gastric Bypass — Laparoscopic Roux-en-Y Gastric Bypass was performed according to the following standards: Gastric pouch was constructed using the lesser curvature of the stomach. A 45mm stapler was initially fired horizontally 2 to 3 cm below the gastroesophageal junction and then 2 o 3 additional fires towards the angle of His and against a 32 French intragastric tube completed the vertical transection. Lengths of the biliopancreatic and alimentary limbs were approximately 50, and 150 cm respectively. An antecolic and antegastric gastrojejunostomy, 1.0 to 1.5 cm in size was hand sewn and the jejuno-jejunostomy was completed in a latero-lateral fashion using one fire of 45 mm lineal stapler with hand sewn closure of the common enterotomy.
Procedure: Omentectomy — After laparoscopic gastric bypass, the greater omentum was divided in the middle from the free edge to the colonic margin using ultrasonic energy. Attachments between the omentum and the transverse colon were dissected. The omentum was detached from the stomach transecting the vessels between the right gastroepiploic vessels and the greater curvature of the stomach. Once the omentum was freed from the stomach, the duodenum and the lower pole of the spleen, it was extracted from the abdominal cavity in a sterile plastic bag.
  Arms: Roux-en-Y Gastric Bypass/Omentectomy

SUMMARY:
The aim of the present study was to evaluate the additional effect of sudden visceral fat reduction by omentectomy on Metabolic Syndrome, acute phase reactants and inflammatory mediators in patients with morbid obesity undergoing Laparoscopic Roux-en-Y Gastric Bypass.

DETAILED DESCRIPTION:
Although weight loss controls Metabolic Syndrome and reduces the level of inflammatory markers in patients with Morbid Obesity, patients may enjoy the benefit achieving metabolic control before significant weight loss occurs.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35 Kg/m2
* Metabolic syndrome diagnosed

Exclusion Criteria:

* Type 1 diabetes
* Uncontrolled type 2 diabetes
* Cirrhosis or active hepatitis
* Pregnancy
* Recent MI or stroke

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-12; Primary Completion 2007-10 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel F Herrrera, MD, PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran

REFERENCES:
- [Derived] Herrera MF, Pantoja JP, Velazquez-Fernandez D, Cabiedes J, Aguilar-Salinas C, Garcia-Garcia E, Rivas A, Villeda C, Hernandez-Ramirez DF, Davila A, Zarain A. Potential additional effect of omentectomy on metabolic syndrome, acute-phase reactants, and inflammatory mediators in grade III obese patients undergoing laparoscopic Roux-en-Y gastric bypass: a randomized trial. Diabetes Care. 2010 Jul;33(7):1413-8. doi: 10.2337/dc09-1833. PMID 20587720

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients from the obesity clinic were recruited from November 2005 to October 2006
Period: Overall Study
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Started | 12 | 12
Completed | 11 (Patient didn't complete the follow-up period after surgery) | 11 (Patient didn't complete the follow-up period after surgery)
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.8 (12.9) | 39.8 (11.1) | 38.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Components of Metabolic Syndrome (Body Mass Index)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
Kg/m2 | 44.9 (3.1) | 44.5 (4.3)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.79, t-test, 2 sided

2. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Interleukine-6)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
pg/ml | 4.8 (9.5) | 8.9 (16.9)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.49, t-test, 2 sided

3. Primary Outcome: Components of Metabolic Syndrome (Body Mass Index)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 month
Measure: Median (Standard Deviation); unit: Kg/m2
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
Kg/m2 | 40.1 (3.0) | 40 (3.9)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.96, t-test, 2 sided

4. Primary Outcome: Components of Metabolic Syndrome (Body Mass Index)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
Kg/m2 | 36.5 (3.0) | 36.2 (3.8)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = .86, t-test, 2 sided

5. Primary Outcome: Components of Metabolic Syndrome (Body Mass Index)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
Kg/m2 | 32.4 (2.9) | 33.2 (3.6)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.60, t-test, 2 sided

6. Primary Outcome: Components of Metabolic Syndrome (Body Mass Index)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
Kg/m2 | 30.3 (2.5) | 30.7 (3.8)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.76, t-test, 2 sided

7. Primary Outcome: Components of Metabolic Syndrome (Systolic Blood Pressure)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mmHg | 131.8 (9.8) | 134.6 (6.9)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.45, t-test, 2 sided

8. Primary Outcome: Components of Metabolic Syndrome (Systolic Blood Pressure)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mmHg | 120 (20) | 116.7 (11.5)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.81, t-test, 2 sided

9. Primary Outcome: Components of Metabolic Syndrome (Systolic Blood Pressure)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mmHg | 115.6 (9.0) | 115 (7.1)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.92, t-test, 2 sided

10. Primary Outcome: Components of Metabolic Syndrome (Systolic Blood Pressure)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mmHg | 108.3 (9.8) | 125 (10.7)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.01, t-test, 2 sided

11. Primary Outcome: Components of Metabolic Syndrome (Systolic Blood Pressure)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mmHg | 116.7 (5.2) | 124.3 (11.4)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.15, t-test, 2 sided

12. Primary Outcome: Components of Metabolic Syndrome (Diastolic Blood Pressure)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mmHg | 85.5 (7.9) | 89 (3.9)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.20, t-test, 2 sided

13. Primary Outcome: Components of Metabolic Syndrome (Diastolic Blood Pressure)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mmHg | 70 (17.3) | 76.7 (15.3)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.64, t-test, 2 sided

14. Primary Outcome: Components of Metabolic Syndrome (Diastolic Blood Pressure)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mmHg | 74.4 (8.2) | 75 (7.1)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.92, t-test, 2 sided

15. Primary Outcome: Components of Metabolic Syndrome (Diastolic Blood Pressure)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mmHg | 70 (6.3) | 81.3 (6.4)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

16. Primary Outcome: Components of Metabolic Syndrome (Diastolic Blood Pressure)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mmHg | 71.7 (4.1) | 76.6 (8.7)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.21, t-test, 2 sided

17. Primary Outcome: Components of Metabolic Syndrome (Glucose)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 99.8 (8.6) | 105 (35.6)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.65, t-test, 2 sided

18. Primary Outcome: Components of Metabolic Syndrome (Glucose)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 96.6 (25.7) | 88.3 (10.8)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.33, t-test, 2 sided

19. Primary Outcome: Components of Metabolic Syndrome (Glucose)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 87.5 (9.4) | 90.5 (5.7)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.39, t-test, 2 sided

20. Primary Outcome: Components of Metabolic Syndrome (Glucose)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 87.6 (4.8) | 85.5 (7.8)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.47, t-test, 2 sided

21. Primary Outcome: Components of Metabolic Syndrome (Glucose)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 88.1 (9.4) | 89.3 (7.9)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.75, t-test, 2 sided

22. Primary Outcome: Components of Metabolic Syndrome (Insulin)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: μU/μL
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
μU/μL | 21.6 (9.8) | 22 (12.4)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.94, t-test, 2 sided

23. Primary Outcome: Components of Metabolic Syndrome (Insulin)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: μU/μL
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
μU/μL | 9.8 (3.0) | 10.4 (4.9)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.74, t-test, 2 sided

24. Primary Outcome: Components of Metabolic Syndrome (Insulin)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: μU/μL
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
μU/μL | 8.4 (2.7) | 7.9 (2.8)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.72, t-test, 2 sided

25. Primary Outcome: Components of Metabolic Syndrome (Insulin)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: μU/μL
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
μU/μL | 7.3 (3.6) | 6.6 (1.5)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.67, t-test, 2 sided

26. Primary Outcome: Components of Metabolic Syndrome (Total Cholesterol)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 182.8 (36.6) | 192.3 (55.4)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.64, t-test, 2 sided

27. Primary Outcome: Components of Metabolic Syndrome (Total Cholesterol)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 125 (22.5) | 159.7 (44.8)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.038, t-test, 2 sided

28. Primary Outcome: Components of Metabolic Syndrome (Total Cholesterol)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 143.4 (29.6) | 167.7 (44.5)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.14, t-test, 2 sided

29. Primary Outcome: Components of Metabolic Syndrome (Total Cholesterol)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 155.2 (27.7) | 171.9 (31.6)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.21, t-test, 2 sided

30. Primary Outcome: Components of Metabolic Syndrome (Total Cholesterol)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 157.4 (25.9) | 166.6 (25.9)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.42, t-test, 2 sided

31. Primary Outcome: Components of Metabolic Syndrome (Triglycerides)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 180.4 (83.8) | 292.4 (248.3)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.18, t-test, 2 sided

32. Primary Outcome: Components of Metabolic Syndrome (Triglycerides)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 108.7 (40.1) | 150.1 (69.2)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.10, t-test, 2 sided

33. Primary Outcome: Components of Metabolic Syndrome (Triglycerides)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 108.6 (36.7) | 140.5 (62.2)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.16, t-test, 2 sided

34. Primary Outcome: Components of Metabolic Syndrome (Triglycerides)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 123.1 (28.3) | 159.3 (79.8)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.18, t-test, 2 sided

35. Primary Outcome: Components of Metabolic Syndrome (Triglycerides)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 99.1 (34) | 118 (62.2)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.40, t-test, 2 sided

36. Primary Outcome: Components of Metabolic Syndrome (Low-Density Lipoproteins)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 106.8 (32.3) | 126.6 (50)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.44, t-test, 2 sided

37. Primary Outcome: Components of Metabolic Syndrome (Low-Density Lipoproteins)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 71.4 (14.7) | 104.2 (43.3)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.035, t-test, 2 sided

38. Primary Outcome: Components of Metabolic Syndrome (Low-Density Lipoproteins)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 77.1 (23.7) | 104.1 (37.6)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.07, t-test, 2 sided

39. Primary Outcome: Components of Metabolic Syndrome (Low-Density Lipoproteins)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 91.1 (21.9) | 91 (32.1)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.99, t-test, 2 sided

40. Primary Outcome: Components of Metabolic Syndrome (Low-Density Lipoproteins)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 95 (18.2) | 94.6 (17.2)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.96, t-test, 2 sided

41. Primary Outcome: Components of Metabolic Syndrome (High-Density Lipoproteins)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 38.6 (9.1) | 35.5 (10.1)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.44, t-test, 2 sided

42. Primary Outcome: Components of Metabolic Syndrome (High-Density Lipoproteins)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 31.5 (9.7) | 31.4 (7.8)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.97, t-test, 2 sided

43. Primary Outcome: Components of Metabolic Syndrome (High-Density Lipoproteins)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 34.8 (10) | 35.5 (8.6)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.85, t-test, 2 sided

44. Primary Outcome: Components of Metabolic Syndrome (High-Density Lipoproteins)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 38.3 (12.5) | 40.9 (10.6)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.61, t-test, 2 sided

45. Primary Outcome: Components of Metabolic Syndrome (High-Density Lipoproteins)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
mg/dl | 42.9 (8.7) | 45.8 (12.8)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.55, t-test, 2 sided

46. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Interleukine-6)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
pg/ml | 17.2 (36.9) | 11.2 (20.6)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.65, t-test, 2 sided

47. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Interleukine-6)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
pg/ml | 9.9 (27.8) | 6.8 (12.3)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.74, t-test, 2 sided

48. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Interleukine-6)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
pg/ml | 4.3 (5.6) | 6.0 (7.2)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.57, t-test, 2 sided

49. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (C-reactive Protein)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
μg/mL | 64.5 (75.4) | 69.2 (57.2)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.87, t-test, 2 sided

50. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (C-reactive Protein)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
μg/mL | 29.6 (35.7) | 16.5 (16.4)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.28, t-test, 2 sided

51. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (C-reactive Protein)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
μg/mL | 22.2 (33.6) | 16.7 (18.4)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy; Test type: Superiority or Other; p = 0.64, t-test, 2 sided

52. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (C-reactive Protein)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
μg/mL | 8.9 (20.1) | 2.8 (3.1)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.42, t-test, 2 sided

53. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Tumor Necrosis Factor-alpha)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
pg/ml | 5.2 (3.3) | 5.7 (2.7)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.72, t-test, 2 sided

54. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Tumor Necrosis Factor-alpha)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
pg/ml | 5.3 (2.3) | 4.9 (1.9)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.68, t-test, 2 sided

55. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Tumor Necrosis Factor-alpha)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
pg/ml | 2.5 (2.6) | 4.7 (2.9)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.08, t-test, 2 sided

56. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Tumor Necrosis Factor-alpha)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
pg/ml | 5.9 (7.1) | 4.8 (3.5)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.71, t-test, 2 sided

57. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Leptin)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
ng/ml | 55.4 (30) | 103.6 (153.1)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.32, t-test, 2 sided

58. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Leptin)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
ng/ml | 39.8 (23.6) | 44.7 (24.4)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.64, t-test, 2 sided

59. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Leptin)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
ng/ml | 52.4 (35.5) | 65.8 (57.9)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.52, t-test, 2 sided

60. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Leptin)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
ng/ml | 55 (39.6) | 87 (57.1)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.59, t-test, 2 sided

61. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Adiponectin)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: Basal
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
ng/ml | 10.7 (5.1) | 9.5 (4.8)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.57, t-test, 2 sided

62. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Adiponectin)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
ng/ml | 13.9 (4.3) | 15.8 (6.2)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.43, t-test, 2 sided

63. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Adiponectin)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
ng/ml | 18.7 (6.6) | 17.7 (6.5)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.72, t-test, 2 sided

64. Secondary Outcome: Acute Phase Reactants and Inflammatory Mediators (Adiponectin)
Description: Absolute values are presented, a basal value is provided in a previous outcome measure to determine the improvement.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Number analyzed (Participants) | 11 | 11
ng/ml | 18.9 (5.1) | 16.4 (10.4)
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass/Omentectomy vs Roux-en-Y Gastric Bypass Alone; Test type: Superiority or Other; p = 0.56, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Roux-en-Y Gastric Bypass/Omentectomy | Roux-en-Y Gastric Bypass Alone
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roux-en-Y Gastric Bypass/Omentectomy (N=12) | Roux-en-Y Gastric Bypass Alone (N=12)
Pancreatic Fistula (Surgical and medical procedures) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
An important limitation of our study is the small number of studied patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes